CLINICAL TRIAL: NCT04754763
Title: A Comparative Study On The Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity: A Randomized Clinical Trial
Brief Title: A Comparative Study On The Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Ather Akber, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAkber
Record Dates: First submitted 2021-01-14; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Dentin-Bonding Agents; Propolis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis (Experimental): Propolis was applied by disposable micro brush on particular sensitive teeth and left undisturbed for 60 seconds to let it dry. Followup was done at 7th, 15th and 30th day
  Interventions: Drug: Propolis
- Seventh generation Dentine Bonding Agent (Scotchbond™ Universal Adhesive, 3M ESPE) (Active Comparator): Application of Seventh generation Dentine Bonding Agent (Scotchbond™ Universal Adhesive, 3M ESPE) on sensitive surfaces was applied single coated for 20 seconds, gently applied air for 5 seconds and cured for 10 seconds (as per manufacturer's instructions). Followup was done at 7th, 15th and 30th day
  Interventions: Drug: Dentin-Bonding Agents

INTERVENTIONS:
Drug: Dentin-Bonding Agents — 3M ESPE Scotchbond™ Universal Adhesive systems is a seventh generation single-bottled one-step self-etch adhesive system.
  Arms: Seventh generation Dentine Bonding Agent (Scotchbond™ Universal Adhesive, 3M ESPE)
Drug: Propolis — Propolis was obtained from Margalla hills, Islamabad by NARC (National Agriculture Research Council, Islamabad). Plant source origin is Acacia modesta and Apis mellifera bees collect it. The 30% ethanolic extract of propolis from raw propolis was obtained in Pakistan Council of Scientific & Industrial Research (PCSIR) by dissolving the propolis in 95% ethanol and straining out the precipitate
  Arms: Propolis

SUMMARY:
Background:

Dentine hypersensitivity (DH) causes considerable pain and discomfort to an individual due to number of stimuli on exposed dentine. Different kinds of treatment strategies are used in the resolution of dentine hypersensitivity including the use of propolis and dentine bonding agent. No study had compared the efficacy of propolis and dentine bonding agent.

Objective:

The objective of the study was to find out whether there is a difference in the efficacy of Propolis and seventh generation dentine bonding agent in reducing the dentine hypersensitivity. Comparison within the groups and pairwise comparisons were also recorded in reducing dentine hypersensitivity.

Methods:

In this six month In- Vivo single blinded randomized clinical study, a total number of 52 patients with complain of dentine hypersensitivity were selected in two groups after taking informed consent. Group A and B received 30% ethanolic extract of propolis and dentine bonding agents respectively by a trained operator. Recordings of dentine hypersensitivity were obtained at Day 0, before and after the application of experimental agents, and also on Day 7, 15 and 30 by the principal investigator. Response was measured by Visual Analog Scale and Schiff Cold Air Sensitivity Scale. Statistical Package for the Social Sciences (SPSS) version 20 was used to analyze the data with level of significance set at p < 0.05. Friedman test was applied to see the comparison within groups and Wilcoxon Signed Rank test was used for Pairwise comparison. Mann Whitney U-Test was applied for comparison between groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients reporting to Periodontology department of Dow International Dental College (DIDC) with dentine hypersensitivity
* Patients having age of 20- 45 years
* Systemically healthy patients
* Patients having at least 2 vital teeth with hypersensitivity
* Patients having sensitivity on facial surfaces to air stimulus
* Patients with Score I of Silness and Loe Plaque Index 77
* Patients who used Fluoride dentifrices for hypersensitivity but could not get relief from it.

Exclusion Criteria:

* Patients with carious, cracked or restored teeth, abutment teeth used of removable or fixed prosthesis and tooth with any other dental pathology
* Patients who used analgesics, mood alteration drugs during last six months
* Smoker, pregnant and nursing mothers
* Patients who used tooth whitening or bleaching agents in the last six months
* Patients who were undergoing orthodontic therapy and history of periodontal surgery during last six months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Before application of experimental agents (Day 0)
  Treatment of dentine hypersensitivity assessed with the help of Visual Analog Scale (VAS). Recordings were obtained at Day 0, before the application of experimental agents.
  Visual Analog Scale which will be scored as 0 (No Pain), 1-3 (Mild Pain), 4-6 (Moderate Pain) and 7-10 (Severe Pain).
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Before application of experimental agents (Day 0)
  Treatment of dentine hypersensitivity assessed with the help of Schiff Cold Air Sensitivity Scale. Recordings were obtained at Day 0, before the application of experimental agents.
  Schiff Cold Air Sensitivity Scale is mainly used to evaluate subject response to a stimulus like air or evaporative. This scale is scored as follows:
  1. Subject does not respond to air stimulus.
  2. Subject responds to air stimulus but does not request discontinuation of stimulus.
  3. Subject responds to air stimulus and requests discontinuation or moves from stimulus.
  4. Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | 1 minute after application of experimental agents (Day 0)
  Treatment of dentine hypersensitivity assessed with the help of Visual Analog Scale (VAS). Scale. Recordings were obtained at Day 0, after the application of experimental agents.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | 1 minute after application of experimental agents (Day 0)
  Treatment of dentine hypersensitivity assessed with the help of Schiff Cold Air Sensitivity Scale. Recordings were obtained at Day 0, after the application of experimental agents.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 7
  Treatment of dentine hypersensitivity assessed with the help of Visual Analog Scale (VAS). Recordings were obtained on Day 7.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 7
  Treatment of dentine hypersensitivity assessed with the help of Schiff Cold Air Sensitivity Scale. Recordings were obtained on Day 7.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 15
  Treatment of dentine hypersensitivity assessed with the help of Visual Analog Scale (VAS). Recordings were obtained on Day 15.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 15
  Treatment of dentine hypersensitivity assessed with the help of Schiff Cold Air Sensitivity Scale. Recordings were obtained on Day 15.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 30
  Treatment of dentine hypersensitivity assessed with the help of Visual Analog Scale (VAS). Recordings were obtained on Day 30.
Effect Of Propolis And Dentine Bonding Agent In Treating Dentine Hypersensitivity | Day 30
  Treatment of dentine hypersensitivity assessed with the help of Schiff Cold Air Sensitivity Scale. Recordings were obtained on Day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Ather Akber, M.Sc, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow International Dental Campus (Defence Campus), Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04754763/Prot_SAP_ICF_000.pdf